CLINICAL TRIAL: NCT01508468
Title: Prospective Randomized Multicentric Open Label Study to Evaluate Rituximab Treatment for Idiopathic Membranous Nephropathy (IMN)
Brief Title: Evaluate Rituximab Treatment for Idiopathic Membranous Nephropathy
Acronym: GEMRITUX
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P 100115; AOM 10089 (Other: Assistance Publique)
Record Dates: First submitted 2011-12-09; First posted 2012-01-12 (Estimated); Last update posted 2021-10-26 (Actual); Status verified 2021-10

CONDITIONS: Idiopathic Membranous Nephropathy
Keywords: Rituximab; membranous nephropathy; anti-PLA2R antibody
MeSH Terms: conditions — Glomerulonephritis, Membranous | interventions — Angiotensin II; Adrenergic beta-Antagonists; Hydroxymethylglutaryl-CoA Reductase Inhibitors; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- active comparator (Active Comparator): Non Immunosuppressive Symptomatic Treatment (NIST). "No specific treatment" Converting Enzyme Inhibitor , Angiotensin II receptor antagonist, Anti-renin, Aldosterone antagonist diuretic, Beta blocker, Calcium inhibitor, statin.
  Interventions: Drug: symptomatic treatment (Converting Enzyme inhibitor, Angiotensin II, Anti-renin, Aldosterone antagonist diuretic, Beta blocker, Calcium inhibitor, statin)
- experimental (Experimental): NIST and Rituximab: 500 Mg and 100Mg in solution to be diluted for IV infusion (Mabthera®)
  Interventions: Drug: experimental (Non Immunosuppressive Symptomatic Treatment (NIST) and Rituximab)

INTERVENTIONS:
Drug: symptomatic treatment (Converting Enzyme inhibitor, Angiotensin II, Anti-renin, Aldosterone antagonist diuretic, Beta blocker, Calcium inhibitor, statin) — Converting Enzyme inhibitor , Angiotensin II receptor antagonist, Anti-renin, Aldosterone antagonist diuretic, Beta blocker, Calcium inhibitor, statin.
  Other Names: symptomatic treatment (no specific)
  Arms: active comparator
Drug: experimental (Non Immunosuppressive Symptomatic Treatment (NIST) and Rituximab) — NIST and IV infusion of Rituximab 375mg/m² at day (1) and day (8)
  Other Names: experimental
  Arms: experimental

SUMMARY:
The Membranous Nephropathy is one of the most common cause of Nephrotic Syndrome of adults. In 2/3 of patients the cause of the disease is idiopathic. This can also be referred to as idiopathic membranous nephropathy (IMN).The most of these patients are treated by non immunosuppressive symptomatic treatment (NIST): antiproteinuric and antihypertensive blocking the rennin-angiotensine system. However, the patients resistant to antiproteinuric treatment risk to develop an end stage renal disease (ESRD).

Rituximab has been recently used in patients suffering of nephrotic syndrome related to IMN in four international studies. Rituximab appears effective and safe in reducing proteinuria in nearly 60% of patients.

The primary outcome of the investigators prospective randomized study is to determine whether or not the Rituximab associated with NIST is more effective than non immunologic symptomatic treatment alone in inducing long term remission of proteinuria.

DETAILED DESCRIPTION:
The IMN exposes patients to severe complications which engage the vital prognosis or Nephrotic Syndrome.

The development of well tolerated and effective pathogenesis linked therapies is needed to treat patients with idiopathic Membranous Nephropathy Rituximab, a monoclonal antibody (mAb) against the CD20 present on B cells, has been recently used in patients suffering of nephrotic syndrome related to IMN in four international studies. Rituximab appears effective and safe in reducing proteinuria in nearly 60% of patients.

However, no randomized controlled study has been published to date.

In a previous study, outcome of 28 patients treated with rituximab for idiopathic MN is analysed. Anti-PLA2R antibodies in serum and PLA2R antigen in kidney biopsy were assessed in 10 and 9 patients.

Proteinuria was significantly decreased by 56%, 62% and 87% at 3 months, 6 months and 12 months. At 6 months, 2 patients achieved full remission and 12 partial remission (overall renal response, 50%). At 12 months (n=23), complete remission was achieved in 6 patients and partial remission in 13 patients (overall renal response, 82,6%). Three patients suffered a relapse of nephrotic proteinuria 27 to 50 months after treatment. Univariate analysis suggested that the degree of renal failure (MDRD < 45/ml/min/1.73 m²) is an independent factor that predicts lack of response to rituximab. Anti-PLA2R antibodies were detected in serum in 10 patients, and PLA2R antigen in immune deposits in 8 of 9 patients. Antibodies became negative in all 5 responsive patients with available follow-up. In this retrospective study, a high rate of remission was achieved at 12 months after treatment.

Our trial is a Prospective randomized multicentric open label study. The 2 arms of the study are : Non Immunosuppressive Symptomatic Treatment (NIST) and Rituximab+ NIST Patients randomized to the Rituximab arm will receive 375 mg/m² on days 1 and 8 (+ NIST). Patients in the control arm will be treated only with Non Immunosuppressive Symptomatic Treatment (NIST).

The duration of participation per patient is 6 months for interventional study. An observational follow-up is performed at M9, M12, M18 & M24 for all patients included in study with lab data collection of test done during usual pathology follow-up.

A part of the diagnosis renal biopsy (performed usually as part of health care) is collected for all patients as for the purpose of central analysis.

Our Primary Outcome Measure is evaluation of efficacy of Rituximab associated with NIST in (IMN) in reducing the rate of proteinuria (patients with persistent urinary protein excretion rate ≥3,5g/24 h and albuminemia < 30g/l ).

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old.
* Idiopathic Membranous nephropathy proved by renal biopsy
* Persistent urinary protein excretion rate ≥3,5g/24 h and albuminemia < 30g/l for at least 6 months with full dose of NIST
* Patient receiving a non immunosuppressive conventional treatment (antiproteinuric and antihypertensive blocking the rennin-angiotensine system, lipid-lowering statin) since at least 6 months.
* Patient has given its written consent
* Patient with social coverage (excepting AME)
* Use of an efficient contraception method for women in childbearing age.

Exclusion Criteria:

* Secondary membranous nephropathy
* Patient already in a clinical trial
* Patient received an immunosuppressive treatment within 3 months before the study
* Patient with chronic renal disease defined by estimated GFR by MDRD formula under 30ml/mn/1,73m²
* Pregnancy and breastfeeding
* HIV infection, HCV and HBV active infection
* Severe or evolving infections.
* Allergy or hypersensitivity to Rituximab or any component

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-01-17 (Actual); Primary Completion 2016-08-31 (Actual); Study Completion 2016-08-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of efficacy of Rituximab associated with Non Immunosuppressive Symptomatic Treatment (NIST) in (IMN) in reducing the rate of proteinuria (patients with persistent urinary protein excretion rate ≥3,5g/24 h and albuminemia < 30g/l ) | 6 months
  Evaluation of efficacy of Rituximab associated with Non Immunosuppressive Symptomatic Treatment (NIST) in (IMN) in reducing the rate of proteniuria

SECONDARY OUTCOMES:
Effect of Rituximab on the progression of chronic renal disease | 6 months
  Effect of Rituximab on the progression of chronic renal disease by measuring :
  * Percentage of proteinuria variation at 6 months
  * Percentage of nephrotic syndrome complication: measuring serum creatinine and glomerular filtration rate (GFR) at 6 months, infections, hydrops, vein thrombosis, arterial thrombosis.
Evaluation of Rituximab tolerance in IMN | 6 months
  Evaluation of Rituximab tolerance in IMN :
  -Percentage of serious allergic reaction after Rituximab infusion "drop in blood pressure and/or bronchospasm"
serologic diagnosis with identification of anti-NEP and anti-PLA2R antibodies in IMN before and after treatment with Rituximab | 6 months
  serologic diagnosis with identification of anti-NEP and anti-PLA2R antibodies in IMN before and after treatment with Rituximab
genetic analysis | 6 months
  genetic analysis Study of the alleles "HLA-DQA1 and PLA2R1" situated respectively on chromosomes 6p21 and 2q24.
Lymphocyte CD19 dosing at month 3 and month 6. | 6 months
  Lymphocyte CD19 dosing at month 3 and month 6.

CONTACTS AND LOCATIONS:
Overall Officials: Karine Dahan, MD, Principal Investigator — Assistance Publique
Locations (1):
- Department of Nephrology , Tenon hospital - APHP, Paris, France

REFERENCES:
- [Derived] von Groote TC, Williams G, Au EH, Chen Y, Mathew AT, Hodson EM, Tunnicliffe DJ. Immunosuppressive treatment for primary membranous nephropathy in adults with nephrotic syndrome. Cochrane Database Syst Rev. 2021 Nov 15;11(11):CD004293. doi: 10.1002/14651858.CD004293.pub4. PMID 34778952
- [Derived] Seitz-Polski B, Dahan K, Debiec H, Rousseau A, Andreani M, Zaghrini C, Ticchioni M, Rosenthal A, Benzaken S, Bernard G, Lambeau G, Ronco P, Esnault VLM. High-Dose Rituximab and Early Remission in PLA2R1-Related Membranous Nephropathy. Clin J Am Soc Nephrol. 2019 Aug 7;14(8):1173-1182. doi: 10.2215/CJN.11791018. Epub 2019 Jul 24. PMID 31340979
- [Derived] Dahan K, Debiec H, Plaisier E, Cachanado M, Rousseau A, Wakselman L, Michel PA, Mihout F, Dussol B, Matignon M, Mousson C, Simon T, Ronco P; GEMRITUX Study Group. Rituximab for Severe Membranous Nephropathy: A 6-Month Trial with Extended Follow-Up. J Am Soc Nephrol. 2017 Jan;28(1):348-358. doi: 10.1681/ASN.2016040449. Epub 2016 Jun 27. PMID 27352623